CLINICAL TRIAL: NCT04281758
Title: Comparison of Plasma Caffeine Concentration After Oral Consumption of Caffeinated Beverages With Varied Bioactive Compounds in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PEP-1913
Record Dates: First submitted 2020-02-19; First posted 2020-02-24 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Plasma Caffeine Concentration
Keywords: caffeine; botanicals; beverage; mood
MeSH Terms: interventions — Beverages

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Beverage types are as similar as possible in terms of taste, aroma and color.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Caffeine beverage (control) (Active Comparator): Flavored still beverage with caffeine 100 mg
  Interventions: Other: Beverage
- Caffeine beverage plus bioactive 1 (Experimental): Flavored still beverage with caffeine 100 mg + quercetin 250 mg
  Interventions: Other: Beverage
- Caffeine beverage plus bioactive 2 (Experimental): Flavored still beverage with caffeine 100 mg + curcumin 80 mg
  Interventions: Other: Beverage
- Caffeine beverage plus bioactive 3 (Experimental): Flavored still beverage with caffeine 100 mg + methylliberine 75 mg
  Interventions: Other: Beverage

INTERVENTIONS:
Other: Beverage — 16 oz (473.2 ml)

SUMMARY:
This is a Phase 1, double blind, randomized, controlled, cross-over trial.

The primary outcome is to quantify the incremental area-under-the-concentration-curve (iAUC) for plasma caffeine after oral consumption of caffeinated beverages with various bioactive compounds vs. caffeine alone, in 16 healthy volunteers

Secondary outcomes are caffeine concentration at each time point from pre-dose baseline to 3.5 hrs post-dose, peak caffeine concentration (Cmax), time to maximum caffeine concentration (Tmax) and return to baseline concentration (TBR) for plasma caffeine

Other outcomes are ratings of physiological symptoms and mood, assessed using visual analog scales (VAS).

Polyphenol food frequency questionnaire data at screening will be collected as a possible co-variate.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male volunteers aged 18 to 55 years.
2. Have a BMI of 18 to 29 kg/m2 (inclusive)
3. Able to comprehend and willing to sign an Informed Consent Form (ICF).
4. Willing to avoid caffeine for ≥48 hrs prior to visits
5. Willing to avoid alcohol for ≥24 hrs prior to visits
6. Willing to fast 10 hrs prior to visits
7. Willing to stick to their usual dietary patterns
8. Willing to stick to their usual physical activity level throughout the study
9. No participation in any clinical trial within the past 30 days or any PEP protocol within the past 6 months.

Exclusion Criteria:

1. Reported history or clinical manifestations of significant metabolic (including type 1 or type 2 diabetes mellitus), hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, urological, neurological, or psychiatric disorders.
2. Current or recent history (<30 days prior to Screening) of a clinically significant bacterial, fungal, or mycobacterial infection
3. Current clinically significant viral infection
4. History of malignancy, with the exception of cured basal cell or squamous cell carcinoma of the skin
5. Resting heart rate less than 45 bpm or greater than 100 bpm.
6. History of unstable ischemic heart disease or uncontrolled hypertension (blood pressure greater than or equal to 150/90 mm Hg)
7. History of stomach or intestinal surgery, except that appendectomy and/or cholecystectomy will be allowed.
8. Presence of a malabsorption syndrome possibly affecting drug/Product absorption (e.g., Crohn's disease or chronic pancreatitis).
9. Extreme dietary habits, including but not limited to vegetarian diets and intentional consumption of a high fiber diet, gluten-free, low-carb, vegan, ketogenic.
10. History of alcoholism or drug addiction within 1 year prior to Screening, or current alcohol or drug use that, in the opinion of the investigator, will interfere with the subject's ability to comply with the dosing schedule and study evaluations.
11. Use of any tobacco-containing or nicotine-containing products (including cigarette, pipe, cigar, chewing tobacco, nicotine patch, or nicotine gum and vaping products) within 2 months prior to study entry.
12. Use of any prescription or nonprescription drugs (including vitamins, minerals, and phytotherapeutic, herbal, or plant-derived preparations) is prohibited within 7 days prior to the dose of study product, unless deemed acceptable by the Investigator.
13. Use of alcohol-containing within 24 hours prior to study entry.
14. Use of caffeine containing products 48 hours prior to each dose of study product and during each dosing day.
15. Donation of blood in excess of 500 ml within 4 weeks prior to study entry or of plasma within 2 weeks prior to Screening.
16. Receipt of blood products within 3 months prior to study entry.
17. Subjects who, in the opinion of the investigator, are unable or unlikely to comply with the dosing schedule and study evaluations

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-13 (Actual)

PRIMARY OUTCOMES:
Incremental area-under-the-concentration-curve (iAUC) | At each of 4 testing days, -30 and 0 min pre-dose, and 15, 30, 45, 60, 90, 120, 150, 180 and 210 minutes post-dose
  Plasma caffeine level

SECONDARY OUTCOMES:
Caffeine concentration | At each of 4 testing days, -30 and 0 min pre-dose, and 15, 30, 45, 60, 90, 120, 150, 180 and 210 minutes post-dose
  Plasma caffeine level
Peak caffeine concentration (Cmax) | At each of 4 testing days, -30 and 0 min pre-dose, and 15, 30, 45, 60, 90, 120, 150, 180 and 210 minutes post-dose
  Plasma caffeine level
Time to maximum concentration (Tmax) | At each of 4 testing days, -30 and 0 min pre-dose, and 15, 30, 45, 60, 90, 120, 150, 180 and 210 minutes post-dose
  Plasma caffeine level
Return to baseline concentration (TBR) | At each of 4 testing days, -30 and 0 min pre-dose, and 15, 30, 45, 60, 90, 120, 150, 180 and 210 minutes post-dose
  Plasma caffeine level
Physiological Symptoms | At each of 4 testing days pre-dose, and 60 min, 120 min, and 210 min post-dose
  VAS scale, 9 terms, each rated on a 100 mm line from "Not at all" to "Extremely'. Example, not at all irritable is better than extremely irritable.
Bond-Lader Mood | At each of 4 testing days pre-dose, and 60 min, 120 min, and 210 min post-dose
  VAS scale,16 terms, each rated on a 100 mm line. Example, relaxed is better than tense.

CONTACTS AND LOCATIONS:
Overall Officials: Trisha R Shamp, PhD, Principal Investigator — Prism Clinical Research
Locations (1):
- Prism Clinical Research, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No